CLINICAL TRIAL: NCT04897269
Title: Effectiveness of Progesterone Supplementation for Women Having Low Progesterone Levels on the Day of Frozen Embryo Transfer
Brief Title: Progesterone Supplementation on Women Having Low Progesterone Levels on Transfer Day
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tu Du Hospital (Other Government)
Responsible Party: Principal Investigator, Le Thi Minh Chau, MD, MMSc, PhD, Head of Infertility department of Tu Du hospital, Tu Du Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 656/BVTD-HDDD
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Assisted Reproductive Technology
Keywords: low progesterone levels; progesterone supplementation; clinical pregnancy

STUDY DESIGN:
Intervention Model Description: Patients who have progesterone levels below 10 ng/mL on the day of embryo transfer will be randomized into 2 groups:
  1. Those who will be supplemented with intramuscular progesterone 50mg per day till day of beta-hcg testing
  2. Those who will continue their regular medications
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): In the control group, the patients will be indicated with standard protocol, micronized progesterone (Cyclogest pessary) 400mg two times per day for 14 days, without any progesterone supplementation. If the beta-hcg test is positive, the patients will be treated with the same protocol and followed till 7 weeks of pregnancy when the fetal heart can be confirmed
- Study group (Experimental): In the interventional group,the patients will be indicated with standard protocol, micronized progesterone (Cyclogest pessary) 400mg x 2 per day for 14 days, supplemented with intramuscular progesterone (Progesterone 25mg/ml) 25 mg x 2 at one time per day for 14 days. If the beta-hcg test is positive, the patients will be treated with the same protocol and followed till 7 weeks of pregnancy when the fetal heart can be confirmed
  Interventions: Procedure: Progesterone supplementation

INTERVENTIONS:
Procedure: Progesterone supplementation — This procedure is to add more progesterone on those who have low progesterone levels on the day of embryo transfer
  Arms: Study group

SUMMARY:
The main objective of this study is to compare clinical pregnancy rates between two groups of women who have progesterone levels below 10 ng/mL on the day of frozen embryo transfer: group 1 (vaginal micronized progesterone supplemented with progesterone intramuscular 50 mg per day) and group 2 (vaginal micronized progesterone with no supplementation)

DETAILED DESCRIPTION:
Trial Design:

Single center, longitudinal, randomized, interventional, controlled, pharmacological study, enrolling women attending clinical Centers of medically assisted reproduction (ART).

The study protocol consists in the record of all the diagnostic and clinical outcome parameters, according to clinical practice, for the following patient cohorts:

* The patients who are undergoing frozen embryo transfers with blastocyst or cleavage stage embryos and have progesterone levels below 10 ng/mL on the day of embryo transfer
* Study groups

  * Group supplemented with progesterone intramuscular 50 mg per day until the day of beta-hcg testing (Intervention group);
  * Group with no supplementation (Control group).

    * Endometrial cycle is started with estradiol valerate dose of 4 mg to 8 mg per day, the patients then are appointed to have ultrasound scan of their endometrium every 3 to 7 days and the dose of estradiol may be increased to 16 mg per day maximum depends on the thickness of endometrium; when their endometrium reach 8 mm or higher and duration of endometrial preparation is ≥ 12 days, the embryo transfer will be planned and transvaginal progesterone are prescribed according to the day of transfer.
    * If this is the first cycle of embryo transfer and she is < 35 years of age, 1 grade 1 embryo is transferred, otherwise 2 embryos are transferred.
    * In the morning of embryo-transferred day, all patients will have their blood tested for progesterone levels, if their levels below 10 ng/mL, they will be recruited into the study and randomized into two groups.
    * In the study group, the patients will be prescribed with intramuscular progesterone supplemetation 50 mg + 800mg vaginal micronized progesterone per day for 14 days, until the day of beta-hcg testing.
    * In the control group, the patients will continue their regular medications (800mg vaginal micronized progesterone per day) until the day of beta-hcg testing without any progesterone supplementation.
    * If the beta-hcg test is positive, the patients will be continued their prescriptions depending on study or control group as mentioned above till 7 weeks of pregnancy when the fetal heart can be confirmed, then the patients will be followed up till 11 - 12 weeks of pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone ART with frozen embryo transfer, blastocyst or cleavaged stage embryo transfer, from 18-45 years of age
* Normal BMI
* HRT for Endometrial preparation in FET cycles

Exclusion Criteria:

* Oocyte donor cycles
* Surrogacy
* IVM
* PGT
* Abnormal Uterine (firbroids 0 -> 3 according to FIGO classification, polyp, adenomyosis, congenital malformation)
* Uterus fibroids type 4,5 (Figo classification) > 4cm
* History of recurrent implantation failure
* Endometrial thickness <7mm on the day of ET
* Cesarean scar defect (isthmocele)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We want to investigate on the pregnancy outcome, therefore only female patients will be recruited
Enrollment: 824 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | week 11 - 14 of pregnancy
  defined as the pregnancy completed 11 - 14 weeks of gestation and having vital fetus

SECONDARY OUTCOMES:
implantation rate | 3 weeks after embryo transfer
  the percentage of embryos which successfully undergo implantation compared to the number of embryos transferred in a given period
Pregnancy rate | 2 weeks after embryo transfer
  beta-hCG test is positive
clinical pregnancy rate | 3 weeks after embryo transfer
  pregnancy when fetal heart can be confirmed

CONTACTS AND LOCATIONS:
Overall Officials: Chau TM Le, Principal Investigator — Department of Infertility, Tu Du Hospital
Locations (1):
- Department of Infertility of Tu Du hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cedrin-Durnerin I, Isnard T, Mahdjoub S, Sonigo C, Seroka A, Comtet M, Herbemont C, Sifer C, Grynberg M. Serum progesterone concentration and live birth rate in frozen-thawed embryo transfers with hormonally prepared endometrium. Reprod Biomed Online. 2019 Mar;38(3):472-480. doi: 10.1016/j.rbmo.2018.11.026. Epub 2019 Jan 5. PMID 30642638
- [Result] Gaggiotti-Marre S, Martinez F, Coll L, Garcia S, Alvarez M, Parriego M, Barri PN, Polyzos N, Coroleu B. Low serum progesterone the day prior to frozen embryo transfer of euploid embryos is associated with significant reduction in live birth rates. Gynecol Endocrinol. 2019 May;35(5):439-442. doi: 10.1080/09513590.2018.1534952. Epub 2018 Dec 26. PMID 30585507
- [Result] Labarta E, Mariani G, Holtmann N, Celada P, Remohi J, Bosch E. Low serum progesterone on the day of embryo transfer is associated with a diminished ongoing pregnancy rate in oocyte donation cycles after artificial endometrial preparation: a prospective study. Hum Reprod. 2017 Dec 1;32(12):2437-2442. doi: 10.1093/humrep/dex316. PMID 29040638
- [Result] Volovsky M, Pakes C, Rozen G, Polyakov A. Do serum progesterone levels on day of embryo transfer influence pregnancy outcomes in artificial frozen-thaw cycles? J Assist Reprod Genet. 2020 May;37(5):1129-1135. doi: 10.1007/s10815-020-01713-w. Epub 2020 Feb 10. PMID 32043182
- [Derived] Le TMC, Duong KT, Nguyen QA, Ong PT, Nguyen THN, Thai TCT, Le QT, Roque M, Alviggi C. Effectiveness of progesterone supplementation in women presenting low progesterone levels on the day of frozen embryo transfer: a randomised controlled trial. BMJ Open. 2022 Feb 23;12(2):e057353. doi: 10.1136/bmjopen-2021-057353. PMID 35197354